CLINICAL TRIAL: NCT03212560
Title: Exercise Capacity, Physical Activity Level and Quality of Life in Newly Diagnosed Hematologic Malignant Patients
Brief Title: Exercise Capacity and Physical Activity Levels in Newly Diagnosed Hematologic Malignant Patients
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Other Study IDs: Gazi University1
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hematologic Malignancies
Keywords: Exercise capacity; Physical activity; Quality of life; Pulmonary functions; Muscle strength; Respiratory muscle strength; Respiratory muscle endurance; Dyspnea; Anxiety; Fatigue
MeSH Terms: conditions — Hematologic Neoplasms; Motor Activity; Dyspnea; Anxiety Disorders; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Newly diagnosed individuals: Newly diagnosed hematologic malignant patients included in the study. Inclusion and exclusion criteria were considered.
- Healthy individuals: Those without chronic disease were included in the study. Inclusion and exclusion criteria were considered.

SUMMARY:
Hematologic malignancies are neoplasms that affect the blood, bone marrow, and lymph nodes. Hematological malignancies are the most common forms of leukemia, lymphoma, and myeloma, with numerous subtypes. The general symptoms of leukemia are fatigue, increased susceptibility to infection, bleeding, and the formation of bruises easily. Typical lymphoma symptoms are night sweats and involuntary weight loss, recurrent fever, fatigue, and itching. Myeloma patients often have bone pain, fatigue, anemia, hypercalcemia or infection symptoms.

Adverse effects of hematologic malignancies and treatments cause abnormality in physical function and quality of life. Treatments such as chemotherapy, radiotherapy and hematopoietic stem cell transplantation, which may have side effects on the body systems are used in early or late period. The most common side effect due to chemotherapy is fatigue. Vomiting, weight loss, anemia, depression, decreased aerobic capacity, loss of muscle strength, decreased physical functioning and deterioration in the quality of life are indirect side effects seen in patients.

In the literature, side effects of hematological malignancies have been investigated after treatment in patients. However, no study investigated exercise capacity, quality of life, physical activity level and pulmonary functions on newly diagnosed hematologic malignant patients. Therefore, the investigators aimed to compare aforementioned outcomes in newly diagnosed hematologic malignant patients and healthy controls.

DETAILED DESCRIPTION:
According to sample size calculation 30 newly diagnosed hematologic malignant patients and 30 healthy individuals will be included. Before treatment submaximal exercise capacity, physical activity, quality of life, pulmonary functions, respiratory and peripheral muscle strength, respiratory muscle endurance, dyspnea and fatigue perception, anxiety and depression will be evaluated. Primary outcome measurements are exercise capacity, physical activity, quality of life, secondary outcomes are respiratory and peripheral muscle strength, respiratory muscle endurance, pulmonary functions, dyspnea and fatigue perception, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed hematological malignant patients
* 18-65 years of age
* under standard medications.

Exclusion Criteria:

* having cognitive disorder,
* orthopedic or neurological disease with a potential to affect functional capacity,
* comorbidities such as asthma, chronic obstructive pulmonary disease (COPD), acute infections or pneumonia,
* problems which may prevent evaluating such as visual problems and mucositis
* having metastasis to any region (bone etc.)
* having acute hemorrhage in the intracranial and / or lung and other areas
* having any contraindication to exercise training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity | first day
  Evaluated using 6-minute walking test
Physical activity | first day
  Evaluated using a metabolic holter
General quality of life | second day
  Evaluated using QOL using European Organization for Research and Treatment of Cancer QOL Questionnaire (EORTCQOL)
Disease-specific quality of life | second day
  The Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu)
FACT | second day
  The Functional Assessment of Cancer Therapy-Anemia (FACT-An)

SECONDARY OUTCOMES:
Pulmonary functions | first day
  Evaluated using spirometer
Muscle strength | second day
  Evaluated using hand-held dynamometer for peripheral muscles (shoulder abduction, shoulder flexion, knee extension, hand grip strength)
Respiratory muscle strength | second day
  Evaluated using mouth pressure device
Respiratory muscle endurance | second day
  Evaluated using respiratory muscle trainer (POWERbreathe)
Fatigue | second day
  Evaluated using Fatigue Severity Scale
Dyspnea | first day
  Evaluated using Modified Medical Research Council Dyspnea scale (MMRC)
Activity dyspnea | first day
  Evaluated using Modified Borg Scale
Anxiety | second day
  Evaluated using Hospital Anxiety and Depression Scale
Depression | second day
  Montgomery-Åsberg Depression Rating Scale
Hospital depression | second day
  Evaluated using Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Çelik, Pt, Study Chair — Research assistant; Meral Boşnak Güçlü, Pt, Phd, Study Director — Associate professor; Zübeyde Nur Özkurt, MD, Phd, Principal Investigator — Associate professor
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=.+Paul+KL.+Rehabilitation+and+exercise+considerations+in+hematologic+malignancies.+Am+J+Phys+Med+Rehabil.+2011%3B+90+(5)%3A+88-94.
- See also: Related Info — http://www.google.com.tr/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=0ahUKEwjd7Kmf993UAhUrKsAKHZ6nBBMQFgghMAA&url=http%3A%2F%2Fwww.leukaemia.org.au%2Fdownload.cfm%3Fdownloadfile%3DB56963F0-EA25-11E4-9CF8005056B60026%26typename%3DdmFile%26fieldname%3Dfilename%26filename%3DLLM-WEB6.pdf&usg=AFQjCNHOUG3dtwum5wS8AZxADxPP9X9IPQ
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Cleeland+CS.+Cancer-related+fatigue%3A+new+directions+for+research.+Cancer.+2001%3B+92+(6+suppl)%3A+1657-1661.